CLINICAL TRIAL: NCT05481593
Title: An Accessible and Inclusive Artificial Intelligence Assisted Chronic Disease Self-Management Telehealth Platform: A Pilot Study
Brief Title: An Accessible and Inclusive Artificial Intelligence Assisted Chronic Disease Self-Management Telehealth Platform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Mohanraj Thirumalai, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB-300009485
Record Dates: First submitted 2022-07-27; First posted 2022-08-01 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Disability Physical; Chronic Condition; Chronic Conditions, Multiple
MeSH Terms: conditions — Chronic Disease; Multiple Chronic Conditions

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Scheduled Coaching Calls & Gamified Rewards (Experimental)
  Interventions: Behavioral: Scheduled Coaching + Gamified Rewards
- No Scheduled Coaching Call & Gamified Rewards (Experimental)
  Interventions: Behavioral: No Scheduled Coaching Calls + Gamified Rewards
- Scheduled Coaching Calls & Independent rewards (No Gamification) (Experimental)
  Interventions: Behavioral: Scheduled Coaching Calls + Independent Rewards
- No Scheduled Coaching Calls & Independent Rewards (No Gamification) (Experimental)
  Interventions: Behavioral: No Scheduled Coaching Calls + Independent rewards

INTERVENTIONS:
Behavioral: Scheduled Coaching + Gamified Rewards — Participants will receive scheduled coaching calls and receive gamified rewards (i.e., earning points over time and converted to monetary gifts)
  Arms: Scheduled Coaching Calls & Gamified Rewards
Behavioral: Scheduled Coaching Calls + Independent Rewards — Participants will receive scheduled coaching calls and receive fixed rewards (i.e., non-increasing)
  Arms: Scheduled Coaching Calls & Independent rewards (No Gamification)
Behavioral: No Scheduled Coaching Calls + Gamified Rewards — Participants will not have scheduled coaching calls and receive gamified rewards (i.e., earning points over time and converted to monetary gifts)
  Arms: No Scheduled Coaching Call & Gamified Rewards
Behavioral: No Scheduled Coaching Calls + Independent rewards — Participants will not have scheduled coaching calls and receive fixed rewards (i.e., non-increasing)
  Arms: No Scheduled Coaching Calls & Independent Rewards (No Gamification)

SUMMARY:
The purpose of this study to pilot test an accessible and inclusive artificial intelligence (AI)-assisted, individualized, family-focused lifestyle modification intervention (AI4CHRON) for health-related quality of life for adults with impaired mobility and chronic medical conditions.

DETAILED DESCRIPTION:
The AI4CHRON study will use a four-arm randomized control trial design. Eligible and consented participants will be assigned to one of four groups: 1) Scheduled coaching calls with gamified rewards, 2) Scheduled coaching calls with rewards independent of gamification, 3) No scheduled coaching calls with gamified rewards, and 4) No scheduled coaching calls with rewards independent of gamification. The active intervention period will be six months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosis of heart disease, chronic lung disease, or Type 2 diabetes
* Living with a permanent physical disability (i.e., spina bifida, multiple sclerosis, stroke,)
* Have the ability to converse in and read English
* Availability of a smartphone or computer

Exclusion Criteria:

* Current enrollment in any structured intervention
* Severe cognitive impairment
* Severe untreated depression in the past 6 months
* Major cardiac event in the past 12 months
* Uncontrolled blood pressure
* Resting tachycardia
* Renal failure
* Severe peripheral neuropathy
* Active treatment for cancer in the past 12 months
* Having both visual and hearing impairments (either of them is fine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Health-related quality-of-life | 24 Weeks
  Enabled version of Short-Form 36 (SF-36E)

SECONDARY OUTCOMES:
Physical activity | 24 weeks
  Godin leisure time exercise questionnaire
Usability | 24 weeks
  System Usability Scale
Usability | 24 weeks
  Health Information Technology Usability Evaluation Scale
Medication adherence | 24 weeks
  Medication adherence rating scale
Medication adherence | 24 weeks
  Turnkey Adherence Strategy Medication Adherence
Self-efficacy for managing depression | 24 weeks
  PROMIS SF v1.0 Emotional Distress-Depression 4a
Self-efficacy for managing psychosocial illness | 24 weeks
  PROMIS SF v1.0 Psychosocial illness impact 8a
Self-efficacy for managing emotions | 24 weeks
  PROMIS SF v1.0 Managing Emotions 4a
Self-efficacy for managing medications | 24 weeks
  PROMIS SF v1.0 Managing Emotions 4a
Self-efficacy for managing social interactions | 24 weeks
  PROMIS SF v1.0 Social Interactions 4a
Physical Activity | 24 weeks
  Measured via data from FitBit device (Minutes)
Physical Activity | 24 weeks
  Measured via data from FitBit device (Steps)
Self-efficacy for managing symptoms | 24 weeks
  PROMIS SF v1.0 Managing Symptoms 4a
Self-efficacy for managing daily activities | 24 weeks
  PROMIS SF v1.0 Managing daily activities 4a
Self-efficacy for managing sleep disturbance | 24 weeks
  PROMIS SF v1.0 Sleep Disturbance 4a
Self-efficacy for managing sleep-related impairments | 24 weeks
  PROMIS SF v1.0 Sleep-related impairment
Dietary Intake | 24 weeks
  Short Healthy Eating Index

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Analytic Code

REFERENCES:
- [Derived] Evans E, Zengul A, Subhash Chilke T, Knight A, Willig A, Cherrington A, Mehta T, Thirumalai M. Telehealth Behavioral Intervention for Chronic Disease Self-Management in Adults With Physical Disabilities (My Health, My Life, My Way): Protocol for Intervention Fidelity and Dashboard Design for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Feb 12;13:e53410. doi: 10.2196/53410. PMID 38345845
- [Derived] Evans E, Zengul A, Knight A, Willig A, Cherrington A, Mehta T, Thirumalai M. Stakeholders' Perspectives, Needs, and Barriers to Self-Management for People With Physical Disabilities Experiencing Chronic Conditions: Focus Group Study. JMIR Rehabil Assist Technol. 2023 Dec 18;10:e43309. doi: 10.2196/43309. PMID 38109170
- [Derived] Evans E, Zengul A, Knight A, Willig A, Cherrington A, Mehta T, Thirumalai M. My Health, My Life, My Way-An Inclusive Web-Based Self-management Program for People With Disabilities Living With Chronic Conditions: Protocol for a Multiphase Optimization Strategy Study. JMIR Res Protoc. 2023 Apr 28;12:e31694. doi: 10.2196/31694. PMID 37115620